CLINICAL TRIAL: NCT02046616
Title: Tocilizumab SC in Patients With Active Rheumatoid Arthritis and Inadequate Response to DMARDs. A Single-Arm, Open-Label Study to Evaluate Safety, Tolerability and Efficacy. In a Subgroup of Patients Inflammation Will Be Measured by Ultrasound.
Brief Title: A Study of Subcutaneous (SC) Tocilizumab (RoActemra/Actemra) in Participants With Active Rheumatoid Arthritis (RA) and Inadequate Response to Disease-Modifying Anti-Rheumatic Drugs (DMARDs)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28691; 2013-002007-34 (EudraCT Number)
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Methotrexate

ARMS (1):
- Tocilizumab Alone or Combined with Methotrexate or Other DMARD (Experimental): All participants will receive tocilizumab as a single fixed dose (monotherapy) or in combination with methotrexate or other non-biologic DMARDs, irrespective of body weight, for 24 weeks.
  Interventions: Drug: Tocilizumab; Drug: Methotrexate; Drug: Non-Biologic DMARDs

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab 162 mg will be administered subcutaneously QW.
  Other Names: RoActemra, Actemra
Drug: Methotrexate — Methotrexate dosing is not specified by the protocol and will be given as per standard practice. Participants must be at a stable dose that was initiated at least 4 weeks prior to baseline.
Drug: Non-Biologic DMARDs — Participants will receive non-biologic DMARDs (same non-biologic DMARD that participant was receiving at time of study entry). Dosing is not specified by the protocol and will be given as per standard practice. Participants must be at a stable dose that was initiated at least 4 weeks prior to baseline.

SUMMARY:
This Phase IIIb, open-label, single-arm study will evaluate the safety, efficacy, and tolerability of SC tocilizumab (RoActemra/Actemra) in monotherapy or in combination with methotrexate or other non-biologic DMARDs in participants with active RA who are naive to tocilizumab. Participants will receive tocilizumab 162 milligrams (mg) subcutaneously weekly (QW) for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Active RA according to the revised ACR (1987) criteria or EULAR/ACR (2010) criteria
* Moderate to severe RA with a DAS28-ESR score >3.2 points
* Inadequate response and/or intolerance to MTX or other non-biologic DMARDs and/or where MTX or other non-biologic DMARDs are inappropriate
* Oral corticosteroids (less than or equal to [</=] 10 mg per day prednisolone or equivalent) and nonsteroidal anti-inflammatory drugs (NSAIDs) permitted if on stable dose regimen for greater than or equal to [>/=] 4 weeks prior to baseline
* Permitted non-biologic DMARDs allowed if at stable dose for >/=4 weeks prior to baseline
* Receiving treatment on an outpatient basis, not including tocilizumab
* Agreement to use reliable means of contraception as defined by protocol, among females of childbearing potential and males with female partners of childbearing potential

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following baseline
* Rheumatic autoimmune disease other than RA
* Functional Class IV as defined by the ACR Classification of Functional Status in Rheumatoid Arthritis
* Diagnosis of juvenile idiopathic arthritis or juvenile RA and/or RA before the age of 16
* Prior history of or current inflammatory joint disease other than RA
* Exposure to tocilizumab or any other biologic DMARDs at any time prior to baseline
* Treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational drug, whichever is longer) of screening
* Intra-articular or parenteral corticosteroids within 4 weeks prior to baseline
* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies
* Evidence of serious concomitant disease or disorder
* Known active current or history of recurrent infection
* Any major episode of infection requiring hospitalization or treatment with intravenous (IV) antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks of screening
* Active tuberculosis requiring treatment within the previous 3 years
* Positive for hepatitis B or hepatitis C
* History of or current active primary or secondary immunodeficiency
* Pregnant or lactating women
* Neuropathies or other conditions that might interfere with pain evaluation
* Inadequate hematologic, renal, or liver function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2014-05-28 (Actual); Primary Completion 2016-09-13 (Actual); Study Completion 2016-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (27):
- Denmark (7):
  - Aalborg Universitetshospital Nord, Reumatologisk Afdeling, Aalborg
  - Glostrup Hospital, Reumatologisk Afdeling, Ambulatoriet, Glostrup Municipality
  - Gentofte Hospital, Medicinsk Afd. C, Klinik for Gigt- og Rygsygdomme, Hellerup
  - Holbæk Sygehus, Medicinsk Afd., Reumatologisk Amb.15-2, Holbæk
  - Sjællands Universitetshospital, Køge; Reumatologisk Afdeling, Køge
  - Odense Universitetshospital, Reumatologisk Afdeling C, Ambulatoriet, Odense
  - Svendborg Sygehus, Reumatologisk Ambulatorium, Svendborg
- Finland (6):
  - Helsinki University Central Hospital; Rheumatology Clinic, Helsinki
  - Kiljavan Lääketutkimus Oy, Hyvinkää
  - Central Hospital of Pohjois-Karjala; Outpatient Clinic of Rheumatology, Joensuu
  - Keski-Suomen Keskussairaala; Sisätautien Klinikka, Jyväskylä
  - Lappeenranta Central Hospital; Outpatient Clinic of Internal Medicine, Lappeenranta
  - Oulu University Hospital; Rheumatology, Oulu
- Norway (5):
  - Ålesund Sykehus; Revmatologisk Avdeling, Ålesund
  - Haukeland Universitetssykehus; Revmatologisk Avdeling, Bergen
  - Drammen sykehus Vestre Viken HF, Revmatologisk avd., Drammen
  - Diakonhjemmet; Reumatolgisk Avdeling, Oslo
  - St. Olavs Hospital; Revmatologisk avdeling, Trondheim
- Sweden (9):
  - Länssjukhuset Ryhov; Ortoped- och Reumatolog kliniken, Jönköping
  - Uni Hospital Linkoeping; Dept. of Rheumatology, Linköping
  - Skånes Universitetssjukhus Lund; Reumatologkliniken, Lund
  - Skånes Universitetssjukhus Malmö; Reumatologkliniken, Malmo
  - Örebro Uni Hospital; Rheumatology, Örebro
  - Simrishamns Sjukhus, Simrishamn
  - Karolinska Sjukhuset; Reumatologkliniken D2-1, Stockholm
  - Akademiska sjukhuset, Reumatologkliniken, Uppsala
  - Västmanlands sjukhus Västerås, Reumatologkliniken, Västerås

REFERENCES:
- [Derived] Hammer HB, Jensen Hansen IM, Jarvinen P, Leirisalo-Repo M, Ziegelasch M, Agular B, Terslev L. Rheumatoid arthritis patients with predominantly tender joints rarely achieve clinical remission despite being in ultrasound remission. Rheumatol Adv Pract. 2021 May 14;5(2):rkab030. doi: 10.1093/rap/rkab030. eCollection 2021. PMID 34131623
- [Derived] Hammer HB, Hansen I, Jarvinen P, Leirisalo-Repo M, Ziegelasch M, Agular B, Terslev L. Major reduction of ultrasound-detected synovitis during subcutaneous tocilizumab treatment: results from a multicentre 24 week study of patients with rheumatoid arthritis. Scand J Rheumatol. 2021 Jul;50(4):262-270. doi: 10.1080/03009742.2020.1845394. Epub 2021 Jan 19. PMID 33464147
- [Derived] Choy E, Caporali R, Xavier R, Fautrel B, Sanmarti R, Bao M, Devenport J, Petho-Schramm A. Effects of concomitant glucocorticoids in TOZURA, a common-framework study programme of subcutaneous tocilizumab in rheumatoid arthritis. Rheumatology (Oxford). 2019 Jun 1;58(6):1056-1064. doi: 10.1093/rheumatology/key393. PMID 30649524
- [Derived] Choy E, Caporali R, Xavier R, Fautrel B, Sanmarti R, Bao M, Bernasconi C, Petho-Schramm A. Subcutaneous tocilizumab in rheumatoid arthritis: findings from the common-framework phase 4 study programme TOZURA conducted in 22 countries. Rheumatology (Oxford). 2018 Mar 1;57(3):499-507. doi: 10.1093/rheumatology/kex443. PMID 29244149

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One hundred thirty-three participants entered the 24-week Treatment Period. Those who completed treatment entered the Follow-Up (FU) Period for an additional 8 weeks.
Groups:
- Tocilizumab Alone or Combined With Methotrexate or Other DMARD: All participants received tocilizumab as a single fixed dose (monotherapy) or in combination with methotrexate or other non-biologic DMARDs at a dose of 162 milligrams (mg), irrespective of body weight, administered subcutaneously weekly (QW) for 24 weeks. An additional 8 weeks were allotted for post-treatment evaluation of safety/immunogenicity.
Period: 24-Week Treatment Period
Arm/Group | Tocilizumab Alone or Combined With Methotrexate or Other DMARD
Started | 133
Completed | 114
Not Completed | 19
Not completed — Anaphylaxis/Serious Hypersensitivity | 1
Not completed — Any Other Adverse Event | 13
Not completed — Insufficient Therapeutic Response | 1
Not completed — Physician Decision | 3
Not completed — Other | 1
Period: 8-Week FU Period
Arm/Group | Tocilizumab Alone or Combined With Methotrexate or Other DMARD
Started | 114
Completed | 113
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Set: all participants who were treated with at least one dose of SC tocilizumab.
Groups:
- Tocilizumab Alone or Combined With Methotrexate or Other DMARD: All participants received tocilizumab as a single fixed dose (monotherapy) or in combination with methotrexate or other non-biologic DMARDs at a dose of 162 mg, irrespective of body weight, administered subcutaneously QW for 24 weeks. An additional 8 weeks were allotted for post-treatment evaluation of safety/immunogenicity.
Arm/Group | Tocilizumab Alone or Combined With Methotrexate or Other DMARD
Number analyzed (Participants) | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Week 12
Description: CDAI was derived as the sum of the following: tender joint count (TJC), swollen joint count (SJC), participant global assessment (PGA) of disease activity, and physician assessment of disease activity. TJC and SJC were taken as the number of tender and swollen joints, respectively, out of 28 assessed joints. PGA and physician assessment of disease activity were scored 0-100 millimeters (mm) and rounded to the nearest centimeter (cm) on a visual analog scale (VAS), where higher scores indicate greater perceived disease activity. The total CDAI score range was 0-76, where higher scores indicate increased disease activity. Change from baseline was averaged among all participants. Negative values indicate improvement/reduction in RA disease activity.
Time Frame: Baseline, Week 12
Population: ITT Set; only those patients who provided data at baseline and at least one post-baseline assessment were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Alone or Combined With Methotrexate or Other DMARD
Number analyzed (Participants) | 133
units on a scale
  Baseline | 24.9 (10.5)
  Change at Week 12: number analyzed (Participants) | 119
  Change at Week 12 | -16.6 (12.1)

2. Secondary Outcome: Change From Baseline in Disease Activity Score 28 (DAS28)-Erythrocyte Sedimentation Rate (ESR) Score
Description: DAS28-ESR was based on TJC, SJC, PGA of disease activity, and laboratory-derived ESR. TJC and SJC were taken as the number of tender and swollen joints, respectively, out of 28 assessed joints. PGA of disease activity was scored 0-100 mm on a VAS, where higher scores indicate greater perceived disease activity. The total DAS28-ESR score was transformed to a single score range of 0-10, where higher scores indicate increased disease activity. Change from baseline was averaged among all participants. Negative values indicate improvement/reduction in RA disease activity.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24
Population: ITT Set; only those patients who provided data at baseline and at least one post-baseline assessment were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Alone or Combined With Methotrexate or Other DMARD
Number analyzed (Participants) | 133
units on a scale
  Baseline | 5.0 (1.1)
  Change at Week 2: number analyzed (Participants) | 127
  Change at Week 2 | -1.4 (1.0)
  Change at Week 4: number analyzed (Participants) | 129
  Change at Week 4 | -2.1 (1.1)
  Change at Week 8: number analyzed (Participants) | 125
  Change at Week 8 | -2.8 (1.3)
  Change at Week 12: number analyzed (Participants) | 119
  Change at Week 12 | -2.9 (1.5)
  Change at Week 16: number analyzed (Participants) | 120
  Change at Week 16 | -3.2 (1.4)
  Change at Week 20: number analyzed (Participants) | 113
  Change at Week 20 | -3.3 (1.4)
  Change at Week 24: number analyzed (Participants) | 114
  Change at Week 24 | -3.3 (1.4)

3. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) Response
Description: ACR response was assessed on the basis of percent improvement (20% for ACR20, 50% for ACR50, 70% for ACR70) in both TJC and SJC as well as at least three of the following: physician assessment of disease activity, PGA of disease activity, PGA of pain, Health Assessment Questionnaire-Disability Index (HAQ-DI), and either ESR or C-reactive protein level. TJC and SJC were taken as the number of tender and swollen joints, out of 68 and 66 assessed joints, respectively. PGA and physician assessments were scored 0-100 mm on a VAS, where higher scores indicate greater perceived disease activity or pain. HAQ-DI was scored using participant responses to 20 questions assessing activities of daily living (ADLs), with total score scale of 0-3, where higher scores indicate increased functional disability. The percentage of participants meeting criteria for each level of ACR response was reported.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24
Population: ITT Set
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Alone or Combined With Methotrexate or Other DMARD
Number analyzed (Participants) | 133
percentage of participants
  ACR20, Week 2: number analyzed (Participants) | 127
  ACR20, Week 2 | 25.2
  ACR20, Week 4: number analyzed (Participants) | 130
  ACR20, Week 4 | 51.5
  ACR20, Week 8: number analyzed (Participants) | 125
  ACR20, Week 8 | 70.4
  ACR20, Week 12: number analyzed (Participants) | 120
  ACR20, Week 12 | 70.8
  ACR20, Week 16: number analyzed (Participants) | 120
  ACR20, Week 16 | 82.5
  ACR20, Week 20: number analyzed (Participants) | 114
  ACR20, Week 20 | 77.2
  ACR20, Week 24: number analyzed (Participants) | 114
  ACR20, Week 24 | 78.1
  ACR50, Week 2: number analyzed (Participants) | 127
  ACR50, Week 2 | 8.7
  ACR50, Week 4: number analyzed (Participants) | 130
  ACR50, Week 4 | 22.3
  ACR50, Week 8: number analyzed (Participants) | 125
  ACR50, Week 8 | 46.4
  ACR50, Week 12 (n=120) | 51.7
  ACR50, Week 16: number analyzed (Participants) | 120
  ACR50, Week 16 | 65.8
  ACR50, Week 20: number analyzed (Participants) | 114
  ACR50, Week 20 | 64.9
  ACR50, Week 24: number analyzed (Participants) | 114
  ACR50, Week 24 | 63.2
  ACR70, Week 2: number analyzed (Participants) | 127
  ACR70, Week 2 | 0.8
  ACR70, Week 4: number analyzed (Participants) | 130
  ACR70, Week 4 | 8.5
  ACR70, Week 8: number analyzed (Participants) | 125
  ACR70, Week 8 | 24.0
  ACR70, Week 12: number analyzed (Participants) | 120
  ACR70, Week 12 | 30.0
  ACR70, Week 16: number analyzed (Participants) | 120
  ACR70, Week 16 | 44.2
  ACR70, Week 20: number analyzed (Participants) | 114
  ACR70, Week 20 | 42.1
  ACR70, Week 24: number analyzed (Participants) | 114
  ACR70, Week 24 | 47.4

4. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Response
Description: EULAR response was assessed by change from baseline and absolute DAS28-ESR score. EULAR response classification was as follows: Good (change >1.2 with absolute score </=3.2), Moderate (change >1.2 with absolute score >3.2 or change >0.6 with absolute score </=5.1), None (change </=0.6 or absolute score >5.1). DAS28-ESR was based on TJC, SJC, and PGA of disease activity, and laboratory-derived ESR. TJC and SJC were taken as the number of tender and swollen joints, respectively, out of 28 assessed joints. PGA of disease activity was scored 0-100 mm on a VAS, where higher scores indicate greater perceived disease activity. The total DAS28-ESR score was transformed to a single score range of 0-10, where higher scores indicate increased disease activity. The percentage of participants meeting criteria for each level of EULAR response was reported.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24
Population: ITT Set
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Alone or Combined With Methotrexate or Other DMARD
Number analyzed (Participants) | 133
percentage of participants
  Week 2, Good: number analyzed (Participants) | 127
  Week 2, Good | 29.1
  Week 2, Moderate: number analyzed (Participants) | 127
  Week 2, Moderate | 47.2
  Week 2, None: number analyzed (Participants) | 127
  Week 2, None | 23.6
  Week 4, Good: number analyzed (Participants) | 129
  Week 4, Good | 51.2
  Week 4, Moderate: number analyzed (Participants) | 129
  Week 4, Moderate | 39.5
  Week 4, None: number analyzed (Participants) | 129
  Week 4, None | 9.3
  Week 8, Good: number analyzed (Participants) | 125
  Week 8, Good | 78.4
  Week 8, Moderate (n=125): number analyzed (Participants) | 125
  Week 8, Moderate (n=125) | 16.8
  Week 8, None: number analyzed (Participants) | 125
  Week 8, None | 4.8
  Week 12, Good (n=119): number analyzed (Participants) | 119
  Week 12, Good (n=119) | 78.2
  Week 12, Moderate: number analyzed (Participants) | 119
  Week 12, Moderate | 16.0
  Week 12, None: number analyzed (Participants) | 119
  Week 12, None | 5.9
  Week 16, Good: number analyzed (Participants) | 120
  Week 16, Good | 87.5
  Week 16, Moderate: number analyzed (Participants) | 120
  Week 16, Moderate | 9.2
  Week 16, None: number analyzed (Participants) | 120
  Week 16, None | 3.3
  Week 20, Good: number analyzed (Participants) | 113
  Week 20, Good | 86.7
  Week 20, Moderate: number analyzed (Participants) | 113
  Week 20, Moderate | 8.8
  Week 20, None: number analyzed (Participants) | 113
  Week 20, None | 4.4
  Week 24, Good: number analyzed (Participants) | 114
  Week 24, Good | 87.7
  Week 24, Moderate: number analyzed (Participants) | 114
  Week 24, Moderate | 9.6
  Week 24, None: number analyzed (Participants) | 114
  Week 24, None | 2.6

5. Secondary Outcome: Change From Baseline in CDAI at Weeks 2, 4, 8, 16, 20, and 24
Description: CDAI was derived as the sum of the following: TJC, SJC, PGA of disease activity, and physician assessment of disease activity. TJC and SJC were taken as the number of tender and swollen joints, respectively, out of 28 assessed joints. PGA and physician assessment of disease activity were scored 0-100 mm and rounded to the nearest cm on a VAS, where higher scores indicate greater perceived disease activity. The total CDAI score range was 0-76, where higher scores indicate increased disease activity. Change from baseline was averaged among all participants. Negative values indicate improvement/reduction in RA disease activity.
Time Frame: Baseline and Weeks 2, 4, 8, 16, 20, 24
Population: ITT Set; only those patients who provided data at baseline and at least one post-baseline assessment were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Alone or Combined With Methotrexate or Other DMARD
Number analyzed (Participants) | 133
units on a scale
  Change at Week 2: number analyzed (Participants) | 126
  Change at Week 2 | -6.2 (8.4)
  Change at Week 4: number analyzed (Participants) | 127
  Change at Week 4 | -10.5 (9.8)
  Change at Week 8: number analyzed (Participants) | 125
  Change at Week 8 | -15.7 (11.0)
  Change at Week 16: number analyzed (Participants) | 120
  Change at Week 16 | -18.8 (11.5)
  Change at Week 20: number analyzed (Participants) | 113
  Change at Week 20 | -18.9 (11.7)
  Change at Week 24: number analyzed (Participants) | 114
  Change at Week 24 | -19.0 (11.7)

6. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI)
Description: SDAI was derived as the sum of the following: TJC, SJC, PGA of disease activity, physician assessment of disease activity, and laboratory-derived C-reactive protein level. TJC and SJC were taken as the number of tender and swollen joints, respectively, out of 28 assessed joints. PGA and physician assessment of disease activity were scored 0-100 mm and rounded to the nearest cm on a VAS, where higher scores indicate greater perceived disease activity. The total SDAI score range was 0-86, where higher scores indicate increased disease activity. Change from baseline was averaged among all participants. Negative values indicate improvement/reduction in RA disease activity.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24
Population: ITT Set; only those patients who provided data at baseline and at least one post-baseline assessment were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Alone or Combined With Methotrexate or Other DMARD
Number analyzed (Participants) | 132
units on a scale
  Baseline | 35.76 (20.71)
  Change at Week 2: number analyzed (Participants) | 124
  Change at Week 2 | -15.37 (16.71)
  Change at Week 4: number analyzed (Participants) | 125
  Change at Week 4 | -20.32 (19.24)
  Change at Week 8: number analyzed (Participants) | 124
  Change at Week 8 | -25.89 (20.88)
  Change at Week 12: number analyzed (Participants) | 119
  Change at Week 12 | -26.19 (23.21)
  Change at Week 16: number analyzed (Participants) | 119
  Change at Week 16 | -29.03 (21.15)
  Change at Week 20: number analyzed (Participants) | 112
  Change at Week 20 | -28.47 (21.26)
  Change at Week 24: number analyzed (Participants) | 113
  Change at Week 24 | -28.93 (20.93)

7. Secondary Outcome: Change From Baseline in TJC
Description: TJC was taken as the number of tender joints out of 28 assessed joints.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24
Population: ITT Set; only those patients who provided data at baseline and at least one post-baseline assessment were analyzed.
Measure: Mean (Standard Deviation); unit: tender joints
Units Other Than Participants: Joints
Arm/Group | Tocilizumab Alone or Combined With Methotrexate or Other DMARD
Number analyzed (Participants) | 133
Number analyzed (Joints) | 28
tender joints
  Baseline | 8.8 (5.2)
  Change at Week 2: number analyzed (Participants) | 127
  Change at Week 2 | -2.1 (5.8)
  Change at Week 4: number analyzed (Participants) | 130
  Change at Week 4 | -3.5 (6.1)
  Change at Week 8: number analyzed (Participants) | 125
  Change at Week 8 | -5.8 (6.3)
  Change at Week 12: number analyzed (Participants) | 120
  Change at Week 12 | -5.5 (7.1)
  Change at Week 16: number analyzed (Participants) | 120
  Change at Week 16 | -6.7 (6.9)
  Change at Week 20: number analyzed (Participants) | 114
  Change at Week 20 | -6.7 (6.5)
  Change at Week 24: number analyzed (Participants) | 114
  Change at Week 24 | -7.1 (5.8)

8. Secondary Outcome: Change From Baseline in SJC
Description: SJC was taken as the number of swollen joints out of 28 assessed joints.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24
Population: ITT Set; only those patients who provided data at baseline and at least one post-baseline assessment were analyzed.
Measure: Mean (Standard Deviation); unit: swollen joints
Units Other Than Participants: Joints
Arm/Group | Tocilizumab Alone or Combined With Methotrexate or Other DMARD
Number analyzed (Participants) | 133
Number analyzed (Joints) | 28
swollen joints
  Baseline | 6.8 (5.5)
  Change at Week 2: number analyzed (Participants) | 127
  Change at Week 2 | -2.3 (4.3)
  Change at Week 4: number analyzed (Participants) | 130
  Change at Week 4 | -3.1 (4.7)
  Change at Week 8: number analyzed (Participants) | 125
  Change at Week 8 | -4.8 (5.1)
  Change at Week 12: number analyzed (Participants) | 120
  Change at Week 12 | -5.3 (5.3)
  Change at Week 16: number analyzed (Participants) | 120
  Change at Week 16 | -5.9 (5.2)
  Change at Week 20: number analyzed (Participants) | 114
  Change at Week 20 | -6.0 (5.4)
  Change at Week 24: number analyzed (Participants) | 114
  Change at Week 24 | -5.4 (5.3)

9. Secondary Outcome: Percentage of Participants With At Least One Adverse Event Leading to Dosage Modification
Description: The percentage of participants with at least one adverse event leading to dose/frequency reduction or temporary dose hold was reported.
Time Frame: Baseline up to Week 24
Population: ITT Set
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Alone or Combined With Methotrexate or Other DMARD
Number analyzed (Participants) | 133
percentage of participants
  Dose/Frequency Reduced Due to Adverse Event | 18.80
  Dose Held Due to Adverse Event | 27.07

10. Secondary Outcome: Number of Participants With Neutralizing Anti-Tocilizumab Antibodies
Description: Participants were evaluated for the presence of anti-tocilizumab antibodies. Confirmatory assays were performed in the case of a positive screen assay result.
Time Frame: Baseline to FU Week 8 (up to 32 weeks overall)
Population: ITT Set
Measure: Number; unit: participants
Arm/Group | Tocilizumab Alone or Combined With Methotrexate or Other DMARD
Number analyzed (Participants) | 132
participants | 1

11. Secondary Outcome: Tocilizumab Concentration
Description: Tocilizumab concentration was determined, averaged among all participants, and expressed in micrograms per milliliter (mcg/mL).
Time Frame: Predose (30 minutes) at baseline; Weeks 12, 24; and FU Week 8 (up to 32 weeks overall)
Population: ITT Set. The Analysis was conducted on those participants with quantifiable tocilizumab concentration at the specified assessment.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Tocilizumab Alone or Combined With Methotrexate or Other DMARD
Number analyzed (Participants) | 133
mcg/mL
  Baseline: number analyzed (Participants) | 3
  Baseline | 0.6 (0.3)
  Week 12: number analyzed (Participants) | 117
  Week 12 | 47.4 (28.1)
  Week 24: number analyzed (Participants) | 112
  Week 24 | 48.0 (27.2)
  FU Week 8: number analyzed (Participants) | 11
  FU Week 8 | 32.8 (19.3)

12. Secondary Outcome: Soluble Interleukin-6 Receptor (sIL-6R) Concentration
Description: sIL-6R concentration was determined, averaged among all participants, and expressed in nanograms per milliliter (ng/mL).
Time Frame: Predose (30 minutes) at baseline; Weeks 12, 24; and FU Week 8 (up to 32 weeks overall)
Population: ITT Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tocilizumab Alone or Combined With Methotrexate or Other DMARD
Number analyzed (Participants) | 133
ng/mL
  Baseline: number analyzed (Participants) | 132
  Baseline | 37.0 (12.7)
  Week 12: number analyzed (Participants) | 120
  Week 12 | 509.4 (138.7)
  Week 24: number analyzed (Participants) | 113
  Week 24 | 520.2 (156.4)
  FU Week 8: number analyzed (Participants) | 36
  FU Week 8 | 166.0 (203.5)

13. Secondary Outcome: Change From Baseline in Patient Global Assessment of Disease Activity According to VAS
Description: PGA of disease activity was scored 0-100 mm on a VAS, where higher scores indicate greater perceived disease activity. Change from baseline was averaged among all participants. Negative values indicate improvement/reduction in RA disease activity.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24
Population: ITT Set; only those patients who provided data at baseline and at least one post-baseline assessment were analyzed.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab Alone or Combined With Methotrexate or Other DMARD
Number analyzed (Participants) | 133
mm
  Baseline | 53.2 (21.1)
  Change at Week 2: number analyzed (Participants) | 128
  Change at Week 2 | -6.8 (18.6)
  Change at Week 4: number analyzed (Participants) | 129
  Change at Week 4 | -20.3 (21.3)
  Change at Week 8: number analyzed (Participants) | 125
  Change at Week 8 | -24.6 (25.8)
  Change at Week 12: number analyzed (Participants) | 119
  Change at Week 12 | -30.3 (25.5)
  Change at Week 16: number analyzed (Participants) | 120
  Change at Week 16 | -32.3 (23.9)
  Change at Week 20: number analyzed (Participants) | 113
  Change at Week 20 | -32.2 (27.1)
  Change at Week 24: number analyzed (Participants) | 114
  Change at Week 24 | -34.3 (24.8)

14. Secondary Outcome: Change From Baseline in Patient Global Assessment of RA-Related Pain According to VAS
Description: PGA of RA-related pain was scored 0-100 mm on a VAS, where higher scores indicate greater perceived pain. Change from baseline was averaged among all participants. Negative values indicate improvement/reduction in RA-related pain.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24
Population: ITT Set; only those patients who provided data at baseline and at least one post-baseline assessment were analyzed.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab Alone or Combined With Methotrexate or Other DMARD
Number analyzed (Participants) | 132
mm
  Baseline | 54.8 (22.1)
  Change at Week 2: number analyzed (Participants) | 126
  Change at Week 2 | -9.1 (20.8)
  Change at Week 4 (n=128): number analyzed (Participants) | 128
  Change at Week 4 (n=128) | -22.5 (24.4)
  Change at Week 8: number analyzed (Participants) | 123
  Change at Week 8 | -28.9 (26.6)
  Change at Week 12: number analyzed (Participants) | 117
  Change at Week 12 | -32.8 (27.5)
  Change at Week 16: number analyzed (Participants) | 118
  Change at Week 16 | -35.6 (25.9)
  Change at Week 20: number analyzed (Participants) | 113
  Change at Week 20 | -35.0 (26.7)
  Change at Week 24: number analyzed (Participants) | 113
  Change at Week 24 | -37.8 (26.3)

15. Secondary Outcome: Change From Baseline in HAQ-DI Score
Description: HAQ-DI consisted of 20 questions assessing ADLs in 8 domains (dress/groom, arise, eat, walk, reach, grip, hygiene) with each item rated 0 (no difficulty) to 3 (unable to do). The highest score recorded for any question in a domain determined the score for that domain, unless assistance was required. The total HAQ-DI score was the sum of domain scores divided by the number of domains answered/scored, for a single score range of 0-3, where higher scores indicate increased functional disability. Change from baseline was averaged among all participants. Negative values indicate improvement in ability to perform ADLs.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24
Population: ITT Set; only those patients who provided data at baseline and at least one post-baseline assessment were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Alone or Combined With Methotrexate or Other DMARD
Number analyzed (Participants) | 133
units on a scale
  Baseline (n=133) | 1.2 (0.6)
  Change at Week 2: number analyzed (Participants) | 128
  Change at Week 2 | -0.1 (0.4)
  Change at Week 4: number analyzed (Participants) | 130
  Change at Week 4 | -0.3 (0.5)
  Change at Week 8: number analyzed (Participants) | 124
  Change at Week 8 | -0.5 (0.5)
  Change at Week 12: number analyzed (Participants) | 119
  Change at Week 12 | -0.5 (0.6)
  Change at Week 16: number analyzed (Participants) | 120
  Change at Week 16 | -0.6 (0.6)
  Change at Week 20: number analyzed (Participants) | 114
  Change at Week 20 | -0.6 (0.6)
  Change at Week 24: number analyzed (Participants) | 114
  Change at Week 24 | -0.6 (0.6)

16. Secondary Outcome: Compliance With Treatment According to Percentage of Injections Administered
Description: Participants were provided with diary cards to record home injections. Compliance with treatment was calculated individually for each participant as the actual number of injections as a percentage of the planned number of injections (up to the point of discontinuation for those who discontinued study treatment prematurely) and then averaged among all participants.
Time Frame: Baseline up to Week 24
Population: ITT Set
Measure: Mean (Standard Deviation); unit: percentage of injections
Arm/Group | Tocilizumab Alone or Combined With Methotrexate or Other DMARD
Number analyzed (Participants) | 133
percentage of injections | 86.78 (23.04) [4.2 to 108.3]

17. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score
Description: FACIT-F consisted of 40 questions/statements assessing chronic illness therapy with special emphasis on fatigue over the past 7 days, with each item rated 0 (not at all) to 4 (very much). During score calculations, negatively-worded item scales (e.g., "I have a lack of energy") were reversed so that higher scores indicated more favorable conditions. The total FACIT-F score was the sum of all item scores and ranged 0-160, and the brief FACIT-F score was the sum of 13 item scores and ranged 0-52, where higher scores indicate greater well-being. Change from baseline was averaged among all participants. Positive values indicate improvement in well-being.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24
Population: ITT Set; only those patients who provided data at baseline and at least one post-baseline assessment were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Alone or Combined With Methotrexate or Other DMARD
Number analyzed (Participants) | 133
units on a scale
  Brief Score, Baseline (n=133) | 32.9 (11.1)
  Brief Score, Change at Week 2: number analyzed (Participants) | 128
  Brief Score, Change at Week 2 | 3.4 (6.9)
  Brief Score, Change at Week 4: number analyzed (Participants) | 130
  Brief Score, Change at Week 4 | 5.7 (8.3)
  Brief Score, Change at Week 8: number analyzed (Participants) | 124
  Brief Score, Change at Week 8 | 6.6 (8.0)
  Brief Score, Change at Week 12: number analyzed (Participants) | 118
  Brief Score, Change at Week 12 | 7.6 (7.8)
  Brief Score, Change at Week 16: number analyzed (Participants) | 120
  Brief Score, Change at Week 16 | 7.9 (9.7)
  Brief Score, Change at Week 20: number analyzed (Participants) | 114
  Brief Score, Change at Week 20 | 8.0 (9.1)
  Brief Score, Change at Week 24: number analyzed (Participants) | 113
  Brief Score, Change at Week 24 | 8.4 (8.5)
  Total Score, Baseline | 106.8 (23.6)
  Total Score, Change at Week 2: number analyzed (Participants) | 128
  Total Score, Change at Week 2 | 6.9 (14.0)
  Total Score, Change at Week 4: number analyzed (Participants) | 129
  Total Score, Change at Week 4 | 13.0 (16.6)
  Total Score, Change at Week 8: number analyzed (Participants) | 124
  Total Score, Change at Week 8 | 15.1 (16.2)
  Total Score, Change at Week 12: number analyzed (Participants) | 118
  Total Score, Change at Week 12 | 17.1 (16.2)
  Total Score, Change at Week 16: number analyzed (Participants) | 118
  Total Score, Change at Week 16 | 18.0 (20.1)
  Total Score, Change at Week 20: number analyzed (Participants) | 114
  Total Score, Change at Week 20 | 18.6 (19.8)
  Total Score, Change at Week 24: number analyzed (Participants) | 111
  Total Score, Change at Week 24 | 20.1 (19.3)

ADVERSE EVENTS:
Time Frame: Baseline up to FU Week 8 (up to 32 weeks overall)
Description: ITT Set
Arm/Group | Tocilizumab Alone or Combined With Methotrexate or Other DMARD
Serious Adverse Events (participants affected / at risk) | 12/133
Other Adverse Events (participants affected / at risk) | 120/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab Alone or Combined With Methotrexate or Other DMARD (N=133)
Acute psychosis (Psychiatric disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 2
Infectious pleural effusion (Infections and infestations) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pneumonia (Infections and infestations) | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transient ischaemic attack (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab Alone or Combined With Methotrexate or Other DMARD (N=133)
Nausea (Gastrointestinal disorders) | 11
Injection site erythema (General disorders) | 7
Nasopharyngitis (Infections and infestations) | 20
Upper respiratory tract infection (Infections and infestations) | 10
Alanine aminotransferase increased (Investigations) | 9
Neutrophil count decreased (Investigations) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 7
Headache (Nervous system disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 10
Hypertension (Vascular disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/ or the publication be postponed in order to protect the Sponsor's intellectual property rights.